CLINICAL TRIAL: NCT04057235
Title: Transforaminal/Posterior Lumbar Interbody Fusion With the FlareHawk® Expandable Interbody Fusion Device: A Retrospective Chart Review Study
Brief Title: Retrospective Review of Integrity Implants FlareHawk® for Lumbar Fusion
Status: Completed | Type: Observational
Sponsor: Integrity Implants Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-00001
Record Dates: First submitted 2019-08-13; First posted 2019-08-15 (Actual); Results first posted 2020-04-14 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: FlareHawk Interbody Fusion System — Expandable lumbar intervertebral body fusion device

SUMMARY:
This is a retrospective clinical study (chart review) of patients who have previously undergone Transforaminal Lumbar Interbody Fusion or Posterior Lumbar Interbody Fusion surgery with the FlareHawk expandable interbody fusion cage at one or two contiguous levels.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the clinical outcomes of patients who have undergone a Transforaminal Lumbar Interbody Fusion (TLIF) or Posterior Lumbar Interbody Fusion (PLIF) procedure with a FlareHawk expandable interbody fusion cage(s) to assess the device's performance and safety when used in accordance with its intended use. The primary hypothesis is that study subjects who received the FlareHawk expandable cage(s) through a TLIF or PLIF procedure experienced fusion by 12 months (+/- 3 mo) follow-up, with improvements in clinical outcomes related to pain and/or disability compared to pre-operative scores. Further, the subjects are hypothesized to have not experienced any unforeseen device- or procedure-related adverse events.

ELIGIBILITY:
Inclusion Criteria:

To be a part of this study, the subject must:

1. Have been at least 18 years of age and skeletally mature at the time of surgery
2. Have had clinical and radiological evidence of degenerative disc disease of the lumbar spine
3. Have been treated with PLIF or TLIF surgery using the FlareHawk expandable interbody cage(s) at 1 or 2 contiguous levels from L2 to S1
4. Have been treated using the FlareHawk expandable interbody fusion cage, according to the approved labeling, between December 1, 2017, and May 31, 2018

Exclusion Criteria:

Subjects must not meet any of the following exclusion criteria to be included in the study:

1. Have a history of fusion surgery at the study level(s) prior to treatment with the FlareHawk device(s)
2. Have had spondylolisthesis unable to be reduced to grade 1 as part of the surgical procedure
3. Have had surgery with the FlareHawk device(s) at more than 2 levels
4. Have had surgery with the FlareHawk device(s) at levels outside the range of L2 to S1
5. Have been treated with any bone grafting material other than autogenous or allogenic bone graft in the FlareHawk device(s) and surrounding disc space
6. Have any contraindications listed in the approved labeling

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of at least 100 patients from at least three sites will be enrolled based on inclusion/exclusion criteria. The retrospective chart review will include the full consecutive series of patients who received TLIF or PLIF surgery using the FlareHawk expandable interbody fusion cage between December 1, 2017, and May 31, 2018. Subjects from that consecutive series will be included in the study based on the pre-defined inclusion and exclusion criteria. All subjects will have been diagnosed with degenerative disc disease of the lumbar spine that required lumbar interbody fusion procedure at one or two levels as per the opinion of the treating surgeon. All subjects who meet the inclusion criteria and do not meet any of the exclusion criteria will be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Domagoj Coric, MD, Principal Investigator — Carolina Neurosurgery & Spine Associates, Charlotte, NC
Locations (3):
- United States (3):
  - Chatham Orthopaedic Associates, Savannah, Georgia
  - Carolina Neurosurgery & Spine Associates, Charlotte, North Carolina
  - Northeast Ohio Spine Center, Akron, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Retrospective Study Arm: Participants who previously underwent Transforaminal Lumbar Interbody Fusion (TLIF) or Posterior Lumbar Interbody Fusion (PLIF) surgery with the FlareHawk® expandable interbody fusion device.
Period: Overall Study
Arm/Group | Single Retrospective Study Arm
Started | 129
Had Radiographic Data | 58
Had ODI Data | 43
Had VAS Back Data | 45
Had VAS Leg Data | 45
Completed | 129 (All 129 participants had data for at least one of the primary/secondary outcomes or adverse events)
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Single Retrospective Study Arm: Participants who previously underwent TLIF or PLIF surgery with the FlareHawk® expandable interbody fusion device.
Arm/Group | Single Retrospective Study Arm
Number analyzed (Participants) | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Gender of one subject not recorded in patient chart
  Participants
    number analyzed (Participants) | 128
    Female | 72
    Male | 56
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 129
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.3 (7.3)
Smoking Status [Count of Participants; unit: Participants] — Population: Smoking status not available for 4 patients
  Participants
    number analyzed (Participants) | 125
    Non-smoker | 73
    Active smoker | 25
    Previous smoker | 27
Co-Morbidities [Count of Participants; unit: Participants]
  Hypertension | 53
  Diabetes | 25
  Obesity (BMI >= 30) | 61
  Hypercholesterolemia | 8
  Coronary Heart Disease | 9
  Hypothyroidism | 6
  Active or History of Cancer | 13
Baseline VAS Leg Pain [Mean (Standard Deviation); unit: units on a scale] — Visual Analog Scale for Leg Pain; Scale = 0-10; 0 = No Pain; 10 = Worst Pain Population: Baseline VAS Leg Pain score was not recorded in patient chart for some subjects
  units on a scale
    number analyzed (Participants) | 53
    (all) | 6.8 (2.9)
Baseline VAS Back Pain [Mean (Standard Deviation); unit: units on a scale] — Visual Analog Scale for Back Pain; Scale = 0-10; 0 = No Pain; 10 = Worst Pain Population: Baseline VAS Back Pain score was not recorded in patient chart for some subjects
  units on a scale
    number analyzed (Participants) | 57
    (all) | 7.7 (2.1)
Baseline ODI [Mean (Standard Deviation); unit: units on a scale] — Oswestry Disability Index; Scale = 0-100
  0-20: Minimal disability 21-40: Moderate Disability 41-60: Severe Disability 61-80: Crippling back pain 81-100: Bed-bound Population: Baseline ODI score was not recorded in patient chart for some subjects
  units on a scale
    number analyzed (Participants) | 56
    (all) | 55.0 (17.5)

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Arthrodesis
Description: Proportion of participants with radiographic arthrodesis at 12 months +/- 3 months as determined using plain radiographic images with assessment based on the Bridwell-Lenke grading system [Bridwell and Lenke et al, 1995].
Time Frame: 12 months +/- 3 months
Population: Participants who had radiographs available at 12 months follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Single Retrospective Study Arm
Number analyzed (Participants) | 58
Participants | 56

2. Secondary Outcome: Change in Visual Analog Scale (VAS) for Leg Pain From Preoperative Baseline to Last Available Follow-up
Description: Visual analog scale for measuring pain intensity related to leg pain. The scale is anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 10).
Time Frame: From baseline to last available follow-up, with an average follow-up of 4.6 ± 4.4 months (range: 0.5-20.5 mo)
Population: Participants who had VAS Leg data available at both baseline and follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Retrospective Study Arm
Number analyzed (Participants) | 45
score on a scale | -3.9 (3.4)

3. Secondary Outcome: Change in Visual Analog Scale (VAS) for Back Pain From Preoperative Baseline to Last Available Follow-up
Description: Visual analog scale for measuring pain intensity related to back pain. The scale is anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 10).
Time Frame: From baseline to last available follow-up, with an average follow-up of 4.4 ± 4.3 months (range: 0.5-20.5 mo)
Population: Participants who had VAS Back data at both baseline and follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Retrospective Study Arm
Number analyzed (Participants) | 45
score on a scale | -3.4 (2.6)

4. Secondary Outcome: Change in Oswestry Disability Index (ODI) From Baseline to Last Available Follow-up
Description: ODI is used to quantify disability related to lower back pain. The final score/index ranges from 0-100. A score of 0-20 reflects minimal disability, 21-40 moderate disability, 41-60 severe disability, 61-80 crippled, and 81-100 bed-bound.
Time Frame: From baseline to last available follow-up, with an average follow-up of 4.4 ± 3.8 months (range: 0.5-20.5 mo)
Population: Participants with both baseline and follow-up ODI data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Retrospective Study Arm
Number analyzed (Participants) | 43
score on a scale | -14.6 (19.1)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at the time of surgery (intraoperative adverse events) and through last patient follow-up, with an average follow-up time of 8.0 ± 4.9 months (range: 0.5-20.5 mo).
Description: Adverse Events were not monitored/assessed with regard to specific Adverse Event Terms.
Arm/Group | Single Retrospective Study Arm
All-Cause Mortality (participants affected / at risk) | 0/129
Serious Adverse Events (participants affected / at risk) | 3/129
Other Adverse Events (participants affected / at risk) | 19/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Retrospective Study Arm (N=129)
Subsequent surgical intervention (Musculoskeletal and connective tissue disorders) | 3 (3) — Revision surgery for failed supplemental instrumentation (pedicle screws or rods; not FlareHawk device) or adjacent segment disease. Adverse Events were not monitored/assessed with regard to specific Adverse Event Terms.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Retrospective Study Arm (N=129)
Mild to Moderate Adverse Events (General disorders) | 19 (22) — Other mild to moderate adverse events commonly associated with lumbar interbody fusion surgery. Adverse Events were not monitored/assessed with regard to specific Adverse Event Terms.

LIMITATIONS AND CAVEATS:
This was a retrospective study of patient chart data. No data was prospectively collected as part of this study. Therefore, follow-up data is limited among the overall cohort.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-15): https://cdn.clinicaltrials.gov/large-docs/35/NCT04057235/Prot_SAP_000.pdf